CLINICAL TRIAL: NCT05154461
Title: Intestinal Ketogenic Inhibition of the Incretin GLP-1
Brief Title: Intestinal Ketone Bodies Interfere With the Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ket001
Record Dates: First submitted 2021-10-08; First posted 2021-12-13 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — Alginates; Pea Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP-1 in relation to the 2 major BHB release sites (Experimental): The magnitude of plasma GLP-1 following an OGTT (75g glucose per os) when beta-hydroxybutyrate (BHB) is released either at an upper gastrointestinal site (alginate encapsulation), or at distal gastrointestinal site (pea-protein encapsulation). BHB is given per-os in a single dose of 18g, plus 2 g encapsulation material; totally 20 g.
  Interventions: Other: Alginate; Other: Pea-protein

INTERVENTIONS:
Other: Alginate — BHB covered in alginate will be realised in stomach-duodenum
Other: Pea-protein — BHB covered in pea-protein will be released in ileum-colon

SUMMARY:
The ketone body (KB) ß-hydroxybutyrate will be given to eight fasting healthy volunteers of both sexes in order to observe the effects after an oral glucose tolerance test (OGTT) over 2 h. Then, a standard lunch will be served at 12.00, as well as an afternoon snack at 15.00. Each participant will be its own control and participates in a randomised two-way cross over design; the KB are released in the stomach-duodenum, or in the ileum-colon. Peripheral blood samples are taken for endpoint GLP-1 analyses.

DETAILED DESCRIPTION:
It has been shown in man that a fatty diet in people with obesity stimulated the release of ketone bodies (KB) in the small intestinal mucosa. This observation was partly explained by an increased level of the ketogenic enzyme 3-hydroxy-3-methylglutaryl-CoA synthase (HMGCS2) in the jejunum of the obese people.

Glucagon-like peptide 1 (GLP-1) is a peptide that is released from the intestinal mucosa and mediates among other things, satiation, as well as insulin-secretion and insulin-sensitivity. In patients with obesity, GLP-1 response to food is attenuated, but it increases following bariatric surgery.

The question arose if the increased KB could be linked to the decreased level of meal-induced GLP-1. Indeed, in mice and rats the increased production of KB could be related to a decreased level of GLP-1. However, such a close relationship has never been shown in man.

The present study tests, therefore, if release of the ketone body beta-hydroxybutyric acid into the intestine on two levels (stomach/duodenum and ileum/colon) of healthy volunteers influences the blood concentration of GLP-1 following an oral glucose tolerance test (OGTT). Glucose, insulin and KB are determined in peripheral plasma according to OGTT-routine.

KB are lipid-derived organic molecules that can serve a circulating energy source during starvation/fasting (or pronged exercise). Beta-hydroxybutyrate (BHB), acetoacetate (AcAc) and acetone ("ketone bodies") are products of acetyl-CoA derived from fatty acids converted to via hepatic mitochondria. The three KB are connected to each by proteolytic interconnection. BHB is the most important source of energy, while AcAc is approximately 25-30% of BHB. Acetone is gas-soluble and is exhaled if ketonemia increases.

The present study utilises ingestion of one KB (BHB) to get an acute, rapid increase in ketonemia. An encapsulation technology is used to differentiate the effect of KB on the small intestine from the effect mainly in the colon. Microcapsules with 1./ alginate, will release the KB in proximal stomach/duodenal intestine, and 2./ pea protein will release in the distal part of the intestine, mainly colon. The microcapsules are of food grade and are produced according to Good Manufacturing Process (GMP) standards (AnaBio Technologies LTD, Cork, Ireland). The KB in the microcapsules will contain 18 g BHB- and Ca+, Mg2+. Together with the encapsulation material (alginate or pea-protein) the total weight will be 20g per dose.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of both sexes
* healthy and without prescribed pharmaceuticals (anticonceptive drugs allowed)
* no symptoms associated with gastrointestinal dysfunction

Exclusion Criteria:

* pregnancy or breastfeeding
* allergy towards standard meals or treatment
* previous substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) of plasma GLP-1 over 120 minutes. | 120 minutes (AUC)
  BHB is given in the upper GI tract (alginate encapsulation) or at the distal GI tract (pea-protein encapsulated). AUC of the plasma GLP-1 concentration (pmol x min) stimulated by an OGTT (75 g glucose per-os given).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Dept of Gastrosurgical R&E, Sahlgrenska Universityhospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Informed Consent Form will be delivered to the study personnel.
Supporting Information: Study Protocol, ICF
Time Frame: From the 12th of October 2021, to end of 2022.
Access Criteria: Laboratory of Surgical Research, Sahlgrenska Universityhospital, Gothenburg, Sweden